CLINICAL TRIAL: NCT04686266
Title: Efficacy of a Virtual Intervention for Informal Caregivers of Adults With Frontotemporal Dementia
Brief Title: Improving Self-Care of Behavioral Variant Frontotemporal Dementia Caregivers
Acronym: ViCCY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 843660
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Behavioral Variant of Frontotemporal Dementia; Caregiver Stress Syndrome
MeSH Terms: conditions — Pick Disease of the Brain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators and all staff involved in collecting assessment data will be blinded to group assignment until after the data are locked. The Health Coaches providing the intervention and the caregiver participants will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ViCCY: Health Information + Health Coaching (Experimental): This group will receive 10 front-loaded sessions of virtual health coaching by trained Health Coaches over 6 months with content based on the theoretical framework our prior research. Sessions are provided using tablets. Initially, sessions are weekly to build the relationship, but the frequency of sessions decreases over time
  Interventions: Behavioral: Health Information + Health Coaching
- Health Information (No Intervention): Caregivers in the Health Information group are asked to spend at least 30 minutes weekly using the computer tablet provided to you by the study team to access recommended websites

INTERVENTIONS:
Behavioral: Health Information + Health Coaching — Virtual Health Coaching for You: The focus of these sessions is helping caregivers take care of themselves. These are virtual health coaching sessions by trained Health Coaches over 6 months with content based on the theoretical framework from our prior research
  Other Names: ViCCY
  Arms: ViCCY: Health Information + Health Coaching

SUMMARY:
The research study is being conducted to evaluate the efficacy of a virtual support intervention to reduce stress and poor self-care for caregivers of persons with behavioral variant Frontotemporal Degeneration (bvFTD) compared to receiving health information alone.

DETAILED DESCRIPTION:
Informal caregivers of persons with Frontotemporal degeneration (FTD) are an understudied population with unique needs. FTD is a common cause of young-onset dementia with no known cure. Behavioral variant FTD (bvFTD) is the most common of the FTD syndromes and involves a progressive disorder of emotional regulation and personality, and significant impairment in executive function. bvFTD caregivers face unique challenges which are particularly stressful, including young age at which the disorder appears, behavioral symptoms like apathy and disinhibition that are severe and appear early in bvFTD, and the lack of appropriate supportive services. Indeed, numerous studies have demonstrated that stress, depression and burden are higher in FTD caregivers than in any of the other ADRDs, yet caregiver interventions tested in specifically in the FTD population have been limited to a few small studies that focus on education around patient behavior management, not caregiver self-care.

The research study is being conducted to evaluate the efficacy of a virtual support intervention to reduce stress and poor self-care for caregivers of persons with behavioral variant Frontotemporal Degeneration (bvFTD) compared to receiving health information alone.

30 caregivers will be randomized 1:1 to a health information: health information + health coaching group. Catered information will be delivered via tablets over 6 months with testing dispersed at baseline, 1 month, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregiver providing care at least 8 hours/week
* Reporting poor self-care on screening (Health Self-Care Neglect Scale, score ≥ 2)
* Able to complete the protocol, e.g., adequate vision and hearing, English speaking
* Caregiver of a patient diagnosed bvFTD

Exclusion Criteria:

* Participation in another support randomized, controlled trial
* Untreated major psychiatric illness (Use of anti-anxiety/anti-depressant medicines is acceptable and will be adjusted in analysis if group imbalance is identified.)
* Caregiver with Cognitive Impairment based on Telephone Interview for Cognitive Status (TICS) score <25

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, School of Nursing, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share the data internally with doctoral students and post-doctoral trainees instead of sharing the data widely with external sources. Internal sharing will allow our trainees to complete meaningful studies using secondary analysis techniques and to finish their programs in a timely fashion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication of our major trial data, we will share data with Penn trainees
Access Criteria: The Principal Investigator will personally review requests from students for use of the data. She will approve requests based on the importance of the questions asked. She will personally oversee progress in analysis and the publication of abstracts and articles based on the data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by clinician referral from the University of Pennsylvania Frontotemporal Degeneration Center between December 2020 to April 2021. The first participant was enrolled in December 2020 and the final was enrolled in April 2021. Data collection began in December 2020 and finished in November 2021.
Pre-assignment Details: Of 43 people contacted for recruitment, 8 declined to participate and 4 were ineligible. 31 were randomized to the protocol.
Period: Overall Study
Arm/Group | ViCCY: Health Information + Health Coaching | Health Information
Started | 15 | 16
Month 1 | 15 | 16
Month 3 | 15 | 15
Month 6 | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant in the Health Information group dropped out at Month 1 and therefore, was removed from all analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | ViCCY: Health Information + Health Coaching | Health Information | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.80 (11.3) | 65.07 (9.95) | 63.93 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race of Caregiver: Black or AA | 1 | 0 | 1
  Race of Caregiver: White or Caucasian | 13 | 13 | 26
  Race of Caregiver: Asian | 0 | 1 | 1
  Race of Caregiver: Other | 0 | 1 | 1
  Race of Caregiver: Multi-Racial | 1 | 0 | 1
Education of Caregiver (years) [Count of Participants; unit: Participants]
  Grade School | 0 | 1 | 1
  High School graduate or GED | 2 | 1 | 3
  Trade School or some college | 1 | 2 | 3
  Bachelor's Degree | 4 | 3 | 7
  Doctoral or Professional Degree | 8 | 8 | 16
Relationship to Patient [Count of Participants; unit: Participants]
  Daughter | 1 | 0 | 1
  Mother | 0 | 1 | 1
  Spouse | 14 | 13 | 27
  Other Relative | 0 | 1 | 1
Time as Caregiver (years) [Mean (Standard Deviation); unit: years] | 4.97 (2.26) | 4.99 (3.26) | 4.98 (2.75)
Clinical Dementia Rating Scale-Frontotemporal Lobar Degeneration (global score) [Mean (Standard Deviation); unit: units on a scale] — The Clinical Dementia Rating Scale-Frontotemporal Lobar Degeneration (CDR-FTLD) is used to characterize several cognitive and functional aspects of dementia including Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care as well as two additional domains, behavior and language. Each section is scored on a scale of 0 to 3 (0 = normal, 0.5 = very mild dementia, 1 = mild dementia, 2 = moderate dementia, 3 = severe dementia). The CDR global score is a weighted algorithm to determine the average score to represent overall impairment.
  units on a scale | 1.82 (0.96) | 1.70 (0.75) | 1.77 (0.85)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Self-Care Inventory (SCI)
Description: 30 items scored 0-100. A higher score indicates better self-care. This theoretically-derived instrument has construct validity. The self-care confidence scale is embedded within this instrument.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ViCCY: Health Information + Health Coaching | Health Information
Number analyzed (Participants) | 15 | 15
score on a scale
  SCI Maintenance Baseline | 71.4 (14.1) | 66.4 (18.3)
  SCI Maintenance Month 6 | 80.4 (12.0) | 68.9 (14.7)
  SCI Management Baseline | 54.6 (21.2) | 56.5 (23.7)
  SCI Management Month 6 | 70.7 (15.6) | 59.4 (26.9)
  SCI Monitoring Baseline | 60.5 (19.8) | 64.6 (25.3)
  SCI Monitoring Month 6 | 77.8 (16.6) | 64.0 (24.4)
  SCI Confidence Baseline | 66.3 (20.1) | 68.1 (22.3)
  SCI Confidence Month 6 | 79.6 (18.7) | 65.3 (23.5)

2. Primary Outcome: Change From Baseline in Frontotemporal Dementia Rating Scale (FTDRS)
Description: The FTDRS includes 30 questions covering 7 categories: behavior, outing and shopping, household chores and telephone, finances, medications, meal preparation and eating, and self care and mobility. Each question is scored on a likert scale of "never" (0) to "all the time (2). Higher scores represents more frequent symptoms. The reported scores are the mean/standard deviation for the first 7 questions (Category: Behavior).
Time Frame: 6 months
Population: skipped question by participant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ViCCY: Health Information + Health Coaching | Health Information
Number analyzed (Participants) | 15 | 15
score on a scale
  Q1- Baseline | 1.67 (0.49) | 1.67 (0.49)
  Q1- Month 6 | 1.93 (0.46) | 1.73 (0.80)
  Q2- Baseline | 1.47 (0.74) | 1.53 (0.64)
  Q2- Month 6 | 1.53 (0.64) | 1.60 (0.83)
  Q3- Baseline: number analyzed (Participants) | 14 | 15
  Q3- Baseline | 2.14 (0.77) | 2.13 (0.52)
  Q3- Month 6 | 2.13 (0.64) | 2.13 (0.52)
  Q4- Baseline | 1.73 (0.70) | 1.80 (0.56)
  Q4- Month 6 | 1.93 (0.46) | 1.93 (0.59)
  Q5- Baseline | 2.00 (0.53) | 1.93 (0.59)
  Q5- Month 6 | 1.93 (0.59) | 1.93 (0.80)
  Q6- Baseline | 1.73 (0.80) | 1.73 (0.46)
  Q6- Month 6 | 1.67 (0.49) | 1.87 (0.74)
  Q7- Baseline | 2.13 (0.92) | 2.00 (0.76)
  Q7- Month 6 | 2.00 (0.76) | 1.93 (0.80)

3. Secondary Outcome: Change From Baseline in Perceived Stress Scale
Description: The Perceived Stress Scale is a 14-item instrument that provides a global rating of an individual's belief in the severity and frequency of stressful experiences during the last month. The Perceived Stress Scale includes 14 items designed to assess symptoms of stress and global measures of the degree of stress experienced in the past month. Each item is scored from 0 (never) to 4 (very often), with total sum scores ranging from 0 to 56; higher scores indicate higher perceived stress.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ViCCY: Health Information + Health Coaching | Health Information
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 23.1 (10.0) | 29.2 (8.7)
  Month 6 | 23.4 (12.4) | 28.4 (8.3)

4. Secondary Outcome: Change From Baseline in Center for Epidemiologic Studies Depression Scale (CES-D)
Description: CES-D is a valid and reliable scale for detecting caregiver depression in dementia. The scoring is on a likert scale 0: Rarely or none of the time (less than 1 day), 1: Some or a little of the time (1-2 days), 2: Occasionally or a moderate amount of time (3-4 days), and 3: Most or all of the time (5-7 days). Higher scores represent greater depressive symptoms. Total scores can range 0 to 60. A score equal or above a 16 means a person is at risk for clinical depression.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ViCCY: Health Information + Health Coaching | Health Information
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 19.7 (15.1) | 19.0 (12.8)
  Month 6 | 15.3 (11.3) | 16.6 (10.4)

5. Secondary Outcome: Change From Baseline in Ways of Coping Questionnaire, Short Form
Description: This 42-item questionnaire measures the use of five different coping styles: avoidance, problem-focused, seeking social support, self-blame, and wishful thinking. The original scale has been used widely since developed by Lazarus in 1985. The short version (30 items) uses a 4-point Likert-scale response format (0 = not used to 3 = used a great deal). Scores range from 0-90 with higher scores indicating greater coping. It is reliable (alpha 0.95) and has construct validity. This instrument has been used numerous times in studies with older adult caregivers.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ViCCY: Health Information + Health Coaching | Health Information
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 22.7 (16.0) | 20.4 (15.0)
  Month 6 | 23.4 (15.9) | 19.1 (14.6)

6. Secondary Outcome: Change From Baseline in Zarit Burden Interview (ZBI)
Description: The ZBI has been used in numerous informal dementia caregiver studies to capture burden associated with providing care to a loved one. Total scores are summed and a range is provided for little to no burden (0-21) to severe burden (61-88).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ViCCY: Health Information + Health Coaching | Health Information
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 38.4 (11.4) | 43.6 (13.6)
  Month 6 | 39.3 (14.9) | 46.3 (12.8)

7. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory
Description: Commonly used scale to evaluate 12 common behaviors in dementia including Delusions, Hallucinations, Agitation/Aggression, Depression, Anxiety, Elation/Euphoria, Apathy/Indifference, Disinhibition, Irritability, Aberrant motor behavior, Sleep and Nighttime Behavior Disorders, Appetite and Eating Disorders. Ratings include the frequency of the occurrence of behaviors (1 = occasionally, 2 = often, 3 = frequently, 4 = very frequently), and the level of severity of behaviors (1 = mild, 2 = moderate, 3 = severe). The behavioral domain total score is the product of the frequency score multiplied by the severity score for that behavior. The NPI total score is the sum of all the individual behavioral domains. Scores range from 0-144. Higher scores demonstrate greater symptoms frequency and severity.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ViCCY: Health Information + Health Coaching | Health Information
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 20.4 (15.7) | 23.4 (17.3)
  Month 6 | 14.6 (8.2) | 23.8 (15.4)

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Arm/Group | ViCCY: Health Information + Health Coaching | Health Information
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
As this was a pilot study, it was not sufficiently powered to observe effects on all dimensions of the Self-Care Inventory or our secondary outcome measures. Our caregivers had a high level of education, which is related to socioeconomic status, and it will be important for future studies to examine other social determinants of health and how that affects self-care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT04686266/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT04686266/ICF_001.pdf